CLINICAL TRIAL: NCT01851577
Title: Engaging Fathers in Home Visitation: Incorporation of a Coparenting Intervention
Brief Title: Engaging Fathers in Home Visitation
Acronym: FF Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CIN001-EngagingFathers; 1R01HD069431-01A1 (NIH)
Record Dates: First submitted 2013-05-07; First posted 2013-05-10 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2018-07

CONDITIONS: Interparental Conflict; Parenting; Parent-child Relations; Fathers
Keywords: Coparenting; Problem solving; Child development; Father involvement
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Foundations coparenting program (Experimental): Family Foundations is a coparenting prevention program that will be administered concurrently with ongoing home visiting.
  Interventions: Behavioral: Family Foundations coparenting program
- Home visiting (Active Comparator): Home visiting "as usual" will be provided without the added Family Foundations coparenting prevention program.
  Interventions: Behavioral: Home visiting

INTERVENTIONS:
Behavioral: Family Foundations coparenting program — Family Foundations is a coparenting program for new mothers and fathers designed to teach them skills needed to parent together effectively and facilitate healthy child development. Family Foundations will be administered concurrently with home visiting.
  Arms: Family Foundations coparenting program
Behavioral: Home visiting — Home visiting is a child abuse prevention approach for new mothers designed to strengthen protective factors and mitigate risk factors in order to promote optimal child development.
  Arms: Home visiting

SUMMARY:
The purpose of this study is to determine the efficacy of Family Foundations that is to be delivered concurrently with home visiting. Delivered prenatally and postnatally, Family Foundations is a coparenting prevention program for new mothers and fathers that is designed to optimize child outcomes by teaching parents how to work together in raising their child. Using a randomized clinical trial design, families will be assigned to receive Family Foundations + home visiting or home visiting alone. A comprehensive assessment is administered at baseline and then at post-intervention, and 9 and 18 months later. It is hypothesized that families receiving Family Foundations will improve in their resolving of conflict from pre-intervention through follow-up. Additional anticipated outcomes are that those receiving the intervention will have more involved fathers, mothers and fathers will report less conflict, and children will have better emotional and behavioral outcomes relative to those who receive home visiting alone.

DETAILED DESCRIPTION:
Home visitation is a prevention program for sociodemographically high risk, first-time mothers and their families that is designed to optimize child health and development. Most home visitation programs seek to engage fathers in the service and promote greater positive involvement with their children, although systematic and efficacious strategies to achieve this have not been developed and tested. Yet, it is well-documented that positive father involvement and mutually supportive relationships between fathers and mothers impart direct benefits to both children and their parents. Building upon previous efforts to incorporate evidence-based interventions into the home visitation setting, this study seeks to adapt Family Foundations, a coparenting intervention with a strong empirical foundation, as an augmented strategy in ongoing home visitation. In a first phase of qualitative investigation, we will adapt the format and content of Family Foundations for implementation in the home, addressing the needs of high risk mothers and fathers, and integrate it into standard home visitation services. In a second phase, a clinical trial will be conducted to determine the efficacy of the adapted intervention (HVFF) in contrast to a control condition of home visitation alone (HVA). Specifically, 300 mother/father dyads in home visitation will be recruited prenatally and randomly assigned to HVFF and HVA conditions. HVFF will consist of 8 in-home and 2 group sessions administered weekly and in two equal parts at approximately 2 months before birth and 4 months postpartum. Both the HVFF and HVA participants will be assessed at pre-intervention, post-intervention (5 months postpartum), and 9 and 18 month follow-ups. A comprehensive assessment battery will be administered at each assessment measuring parental cooperation, quality of parental relationship, father involvement, beliefs about parenting, parental psychological adjustment, and intimate partner violence. After the child's birth, child development and social/emotional adjustment will be measured and parenting practices will be videotaped and subsequently rated for parenting quality. It is hypothesized that, relative to controls, fathers in the HVFF condition will participate more frequently and more positively in standard home visits and will be more involved with their children; mothers and fathers in the HVFF condition will have higher levels of coparenting, and lower levels of depression, parental stress, and child abuse potential; and children in the HVFF condition will be more behaviorally and emotionally well-adjusted. Mediators of intervention outcomes will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* First time, prenatal mother participating in a home visiting program
* Biological father interested in being involved with child
* 18 years of age or older
* English speaking

Exclusion Criteria:

* Current substance dependence
* Current psychosis
* Current intimate partner violence

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2013-05; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
mother and father resolving of conflict | pre-intervention, post-intervention (up to 9 months after pre-intervention), up to 18 months after pre-intervention, up to 27 months after pre-intervention
  Mothers and fathers complete measures of conflict resolution, co-parenting, and problem-solving that reflect their ability to successfully resolve conflict.

SECONDARY OUTCOMES:
child development | post-intervention (up to 9 months after pre-intervention), up to 18 months after pre-intervention, up to 27 months after pre-intervention
  Children are on track developmentally at each assessment point

OTHER OUTCOMES:
father involvement in raising child | pre-intervention, post-intervention (up to 9 months after pre-intervention), up to 18 months after pre-intervention, up to 27 months after pre-intervention
  Fathers are actively involved in their child's life and have a decision-making role as measured by self-report and report by mothers at each assessment point.

CONTACTS AND LOCATIONS:
Overall Officials: Robert T. Ammerman, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Solmeyer AR, Feinberg ME, Coffman DL, Jones DE. The effects of the family foundations prevention program on coparenting and child adjustment: a mediation analysis. Prev Sci. 2014 Apr;15(2):213-223. doi: 10.1007/s11121-013-0366-x. PMID 23404669
- [Background] Feinberg ME, Jones DE, Kan ML, Goslin MC. Effects of family foundations on parents and children: 3.5 years after baseline. J Fam Psychol. 2010 Oct;24(5):532-42. doi: 10.1037/a0020837. PMID 20954763
- [Background] Ammerman RT, Putnam FW, Kopke JE, Gannon TA, Short JA, Van Ginkel JB, Clark MJ, Carrozza MA, Spector AR. Development and implementation of a quality assurance infrastructure in a multisite home visitation program in Ohio and Kentucky. J Prev Interv Community. 2007;34(1-2):89-107. doi: 10.1300/J005v34n01_05. PMID 17890195
- [Derived] Ammerman RT, Peugh JL, Teeters AR, Sakuma KK, Jones DE, Hostetler ML, Van Ginkel JB, Feinberg ME. Promoting parenting in home visiting: A CACE analysis of Family Foundations. J Fam Psychol. 2022 Mar;36(2):225-235. doi: 10.1037/fam0000888. Epub 2021 Jun 24. PMID 34166030
- See also: The FF Project is implemented in Every Child Succeeds, a regional home visiting program. — http://www.everychildsucceeds.org